CLINICAL TRIAL: NCT06133530
Title: Effects of Human Milk Oligosaccharides (HMOs) on Gut Microbiota, Immune System and Metabolism in Adults Wintering Over in Antarctica
Brief Title: Human Milk Oligosaccharides (HMOs) and Gut Microbiota, Immune System in Antarctica
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: IU University of Applied Sciences (Other)
Collaborators: University of Bologna (Other); University of Bonn (Other); National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); University of Lorraine (Other); German Institute of Food Technologies (Unknown); Chr Hansen (Industry); European Space Agency (Other); MVZ Institute for Microecology (Unknown); DLR German Aerospace Center (Other)
Responsible Party: Principal Investigator, Martina Heer, Program Direction Nutritional Sciences, IU University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PreGlu
Record Dates: First submitted 2023-09-25; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Healthy Adults; High Altitude; Isolation, Social
Keywords: Immune status; Isolation; High altitude; Glucose tolerance; Gut microbiota; Short chain fatty acids; Bone turnover markers
MeSH Terms: conditions — Altitude Sickness; Social Isolation | interventions — Maltose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maltose (Placebo Comparator): The placebo contains maltose powder applied orally.
  Interventions: Dietary Supplement: Maltose
- Human milk oligosaccahride (Experimental): The experimental group HMO powder applied orally.
  Interventions: Dietary Supplement: Human milk oligosaccharides

INTERVENTIONS:
Dietary Supplement: Human milk oligosaccharides — Prebiotic
  Arms: Human milk oligosaccahride
Dietary Supplement: Maltose — Control
  Arms: Maltose

SUMMARY:
Human milk oligosaccharides (HMOs) are the third-most abundant component in mothers' milk and are an important prebiotic factor for the development of the gut microbiota of infants, promoting the growth of certain beneficial bacterial strains and providing protection against many bacterial and viral infections. HMOs induce immunomodulatory activity by affecting immune cell populations and functions. In a simulator of the adult human intestinal microbial ecosystem, fermentation of HMOs led to an increase of bifidobacteria in parallel with an increase in short-chain fatty acids as well as a reduction in inflammation markers, supporting the potential of HMOs to provide health benefits also in adults. Long-term stay in microgravity induces many physiological responses, including diminished immune function and impaired glucose tolerance which may lead to rather severe consequences. Similarly, hypoxia conditions as in the Concordia station, affects the immune system and may lead to impaired glucose tolerance and insulin resistance. The hypothesis is that HMOs as a prebiotic supplement will mitigate changes in immune function, glucose tolerance, lipid homeostasis, and neurotransmitter production. It is expected that HMO supplementation will

* Modulate gut microbiota composition and function
* Improve inflammation status
* Improve immune function
* Improve glucose tolerance
* Improve nutritional status
* Prevent changes in neurotransmitters associated with anxiety and depression. During the stay in Antarctica an HMO blend will be supplemented to the verum group of volunteers. The control group will receive a placebo. Experiment days with blood drawing, an oral glucose tolerance test, saliva sampling, and feces samples are planned once before, about every second month in Concordia, and once after return.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of supplementation with prebiotics, a specific mixture of carbohydrates found in breast milk (HMOs), as a measure to improve intestinal flora, inflammatory processes in the gut, general immune status, carbohydrate regulation, fat and bone metabolism and neurological changes in Antarctica. The approximately one-year stay at Concordia Station (Antarctica) at an altitude of about 3200 m includes a long journey and subsequent extreme environmental conditions as well as corresponding adaptation mechanisms and is therefore a very good terrestrial model (analogue model) for investigating changes during space stays. Long-term (i.e. > 6 months) exposure to microgravity leads to numerous physiological responses, including impaired glucose tolerance, reduced immune function and bone loss, which can lead to quite severe health consequences. In this analogue model, similar changes, albeit less severe, are observed with regard to the immune system or glucose tolerance as in space flight.

The composition of the diet significantly influences the composition of the intestinal flora. In particular, dietary carbohydrates provide the substrate for certain bacteria that could have a positive effect on health. Prebiotics are defined as substrates that are selectively used by host microorganisms and that provide health benefits. Prebiotics are digested only by gut microorganisms and stimulate the growth or activity of bacteria in the gut that have shown health benefits or improved well-being. The main nutrients for bacterial growth are non-digestible carbohydrates, which by definition are not digested by the host, in this case the human organism (host). Non-digestible carbohydrates include, for example, resistant starch and dextrins, non-starch polysaccharides (NSPs) (e.g. pectins) and non-digestible oligosaccharides (e.g. Raffinose, inulin, etc.). These carbohydrates are fermented by the intestinal bacteria to short-chain fatty acids (SCFAs), mainly acetic acid, propionic acid and butyric acid. This process takes place mainly in the large intestine, but also in the small intestine. SCFAs are rapidly absorbed by the mucosa of the large intestine and exert whole-body effects, contributing, for example, to the host's energy needs or mediating gut-brain communication, which has a major impact on the physiology and health of the host.

HMOs are also prebiotics and are the third most abundant solid component in breast milk. Most of the research published to date on the effects of HMOs has therefore been conducted on infants. HMOs are not digested in the intestine and are mainly utilised in the large intestine by the bacteria that reside there. In infants, it has been shown that HMOs not only promote a healthy composition of the intestinal flora, but also impair the growth of pathogens and modulate the expression of genes involved in inflammation. Several in vitro and in vivo studies have shown antiviral properties of HMOs against various viruses such as rotavirus, norovirus, HIV and influenza. HMOs play a significant role in the immune system by enhancing the immune response. Initial applications of HMOs in adults have supported these findings.

Therefore, this study aims to investigate how daily administration of 5.5 g of an HMO mixture during hibernation at Concordia Station in Antarctica affects:

* glucose tolerance
* inflammatory processes
* immune function
* fat and bone metabolism and
* Well-being

Study procedure This is a so-called placebo-controlled, randomised intervention study in parallel design. This means that subjects will be randomly selected to receive either the mixture of HMOs daily or a placebo. The study duration for a test person is approx. 20 months. It is divided into an examination phase before departure to Antarctica, approximately in September of a year, six phases during the wintering in Antarctica and one phase approximately 6 months after return.

Each individual phase is identical, one example shown in Figure 1.

Day 1 (Weekend day) Day 2 Day 3 Day 4 Day 5 Fasting blood collection X Oral glucose tolerance-test X Saliva sample X Feces sample X X X (X) Diet log X X X HMO supplementation Daily, onset after first session at Concordia

Figure 1: Representation of each phase (U as in figure 1) of testing

Intervention The intervention, i.e. the treatment measure used in this study, in one group is the daily administration of 5.5 g of a carbohydrate mixture analogous to human milk but produced by bacteria. This amount is certified by the European Control Authority as safe for human consumption. The other group receives a corresponding placebo, Maltose.

Measurement method Blood test and venous access Blood sampling from the peripheral vein is associated with the usual risks of venipuncture. These are haematomas or infections at the puncture site. When a peripheral venous access is placed, in rare cases there may be injuries to the vein (sclerotherapy) and the peripheric nerves. Blood collection and venous access are performed by an experienced doctor, which minimises the risk.

Fasting blood collections Fasting blood samples for analysis of various blood parameters are taken on the same day as the oral glucose tolerance test (OGTT) (see figure 1). Since several blood samples are taken for the OGTT, also after the drink has been taken, a venous access in the form of an indwelling venous cannula (small plastic tube) will be placed in the area of the forearm in order to avoid repeated puncturing of the arm veins.

Glucose tolerance by means of an oral glucose tolerance test The so-called oral glucose tolerance test (OGTT) can be used to determine differences in glucose metabolism (sugar metabolism) between the intervention and control phases. On approximately day 3 of each study phase, a drink will be consumed in the morning, fasting state, which is prepared from 75 g glucose (Medicalfox Gluko 75 powder) and 300 ml drinking water. Blood is taken every 15 minutes in the first hour after the drink is given, and every 30 minutes in the second hour.

Saliva sample Saliva samples will be taken to test certain hormones that reflect stress levels, as well as the reactivity of certain viruses (herpes virus, rotavirus). For this purpose, a small cotton wool roll from a prepared container (salivette) is chewed in the mouth for several minutes and returned to the collection tube once during the examination phase. The saliva obtained is frozen and later analysed in the laboratory.

Faecal collection In order to examine the changes in the intestinal flora, faeces samples are taken on 3 consecutive days in each phase. For this purpose, a so-called 'Feces Catcher' is placed over the toilet to better collect the faeces. Three samples are then taken from these faeces in 3 different tubes. The small spoon in each tube is filled with faeces, put back into the tube, closed and frozen.

Documentation of the diet In order to be able to estimate the influence of the food composition on the intestinal flora, the food consumed is documented on 2 working days and one weekend day. This is done in a prepared dietlog.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy subjects
* Volunteers that are able and declare their willingness to participate in the entire study
* Fasting blood glucose concentration: <120 mg/dL
* Willing to be assigned randomly either to the treatment or the control group
* Successfully pass the medical screening
* Signed informed consent
* Social insurance

Exclusion Criteria:

* Medication that may interfere with the interpretation of the results
* Recent sub-standard nutritional status
* Abuse of drugs, medicine or alcohol
* Participation in another study up to two months before study onset
* Cannot clear a criminal background check
* No signed consent form before the onset of the experiment
* Blood donors in the past three months before the onset of the experiment
* Vegetarian and Vegans

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Area under the serum glucose concentration curve (2 hours) over time
Insulin resistance | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Area under the serum insulin concentration curve (2 hours) over time

SECONDARY OUTCOMES:
Fecal calprotectin | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Concentration changes in feces (µg/g) over time
Fecal zonulin | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Concentration changes in feces (ng/ml) over time
Fecal short chain fatty acids | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Concentration changes in feces (mmol/l) over time
Gut microbiota profiling | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Feces feces will be analyzed for microbiota composition by 16S rRNA gene-based next-generation sequencing; Alpha and beta diversity, taxonomic assignment and relative abundance of bacterial groups will be characterized by bioinformatics.
Saliva cortisol | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Cortisol concentration changes in saliva over time
Saliva DHEA | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  DHEA concentration changes in saliva over time
Inflammation markers in blood | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in blood cytokines concentration (EGF, FGF-2, Eotaxin, TGF-α, G-CSF, Flt-3L, GM-CSF, Fractalkine, IFNa2, IFNy, GRO, IL-10, MCP-3), IL-12P40, MDC, IL-12P70, IL-13, IL-15, sCD40L, IL-17, IL-1RA, IL-1α, IL-9, IL-1β, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IP-10, MCP-1, MIP-1α, MIP-1β, TNFα, TNFβ, VEGF, PDGF-AA, PDGFAB-BB, RANTES) pg/ml changes over time
CRP changes in blood | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes (mg/L) in blood C-reactive protein concentrations over time
Lipid metabolism | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Serum concentration changes of triglycerides, total-, HDL-, LDL-cholesterol over time
Glycated albumin | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Serum concentration changes of blood glycated albumin over time in g/l and %
GLP-1 | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Serum concentration changes of GLP-1 (pmol/l) over time
Fetuin-A | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Serum concentration changes of Fetuin-A (µg/ml) over time

OTHER OUTCOMES:
Viral activation | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Latent herpes virus shedding changes over time
Vitamin D status | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Serum concentration changes of 25-OH and 1,25 OH vitamin D over time
GABA and BDNF | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in serum concentrations of GABA and BDNF (pg/ml) over time
Serotonin in blood | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in serum concentrations of serotonin (ng/ml) over time
Kynurenine in blood | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in serum concentrations of Kynurenine (µmol/l) over time
Changes in further tryptophan metabolites | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in serum concentrations of Kynurenic acid, Quinolinic acid, Picolinic acid, Methylnicotinamide, Quinaldic acid, 3-hydroxykynurenine, Anthranilic acid, Nicotinamide (nmol/l) over time
Bone formation marker | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in serum concentrations of PINP in µg/L
Bone resorption marker | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in serum concentrations of ß-CTX in ng/L
Body weight | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Changes in body weight (kg) over time
Body height | pre-Antarctica
  Measurement of body height to derive changes in body mass index
Profile of mood states | 5 consecutive days at baseline, pre-Antarctica; 5 consecutive days every month during the 12 month stay at Antarctica; 5 consecutive days 6-7 month after return from Antarctica
  The profile of mood states is a psychological rating scale to measure changes in six different dimensions of mood (tension, depression, anger, vigour, fatigue, confusion) measured by a questionnaire. It is a five point scale ranging from "not at all" to "extremely".
Positive and negative affect schedule | 5 consecutive days at baseline, pre-Antarctica; 5 consecutive days every month during the 12 month stay at Antarctica; 5 consecutive days 6-7 month after return from Antarctica
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).
Appraisal of life events scale | baseline, pre-Antarctica; about 6-7 month after return from Antarctica
  The Appraisal of life events scale (ALE) measures three factors of appraisal: threat, challenge and loss. It is an adjective check list of 16 adjectives rated on a 6-point scale (1 = disagree very strongly, 6= agree very strongly) that can be used to assess appraisals of retrospectively recalled stressful events as well as ongoing stressful encounters.
Subjective assessment of performance by a Visual Analogue Scale | baseline, pre-Antarctica; every month during the 12 month stay at Antarctica; about 6-7 month after return from Antarctica
  The subjective Assessment of Performance Visual Analogue Scale measures factors such as stress, pain, and anxiety using a visual analog scale. The scale is a numerical rating scale ranking the respective factors from 1 to 10. A higher score indicates greater intensity of the respective factor.
General health Questionnaire (GHQ) | baseline, pre-Antarctica; every month during the 12 month stay at Antarctica; about 6-7 month after return from Antarctica
  The General health Questionnaire (GHQ) focuses on two major areas - the inability to carry out normal functions and the appearance of new and distressing phenomena. It is a 28 item questionnaire and assesses the respondent's current state and asks if that differs from his or her usual state. Each item is accompanied by four possible responses, typically being 'not at all', 'no more than usual', 'rather more than usual' and 'much more than usual', scoring from 0 to 3, respectively.
Global Physical Activity Questionnaire | baseline, pre-Antarctica
  The Global Physical Activity Questionnaire (GPAQ) comprises 19 questions grouped to capture physical activity undertaken in different behavioral domains: work, transport, discretionary and time spent in sedentary activities. It asks for whether at all and if, how many days and how long the respective activity will usually be carried out.
Depression symptoms | Mid-term of the 12 month stay in Antarctica
  Center for Epidemiologic Studies Depression Scale is a 20-item measure that asks the test subjects to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Nutrient intake | baseline, pre-Antarctica; every 1-2 month from month 4 to 10 during the stay in Antarctica (total stay about 12 month); about 6-7 month after return from Antarctica
  Food frequency questionnaire measuring food habits and dietary intake during 3 consecutive days including one weekend day.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Heer, PhD, Principal Investigator — IU International University of Applied Sciences, Erfurt, Germany
Locations (1):
- IU International University of Applied Sciences, Erfurt, Germany